CLINICAL TRIAL: NCT05977673
Title: Efficacy and Safety of Frontline Tislelizumab in Patients With de Novo Hodgkin Lymphoma Unsuitable for Standard Frontline Chemotherapy: a Phase II, Open-label Study
Brief Title: Efficacy and Safety of Frontline Tislelizumab in Patients With de Novo Hodgkin Lymphoma Unsuitable for Standard Frontline Chemotherapy
Acronym: FIL_Tisle-HL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_Tisle-HL
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hodgkin Lymphoma
Keywords: Lymphoma; Hodgkin; Tislelizumab; PD1; Checkpoint; Inhibitor; De novo; Unsuitable; Chemotherapy; Immune
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab (Experimental): Tislelizumab single dose every 3 weeks up to 35 total administration
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg IV day1

SUMMARY:
This is a multicenter, prospective, non-randomized, open-label, phase 2 clinical study to evaluate the efficacy and safety of tislelizumab in patients with de novo Hodgkin Lymphoma deemed ineligible to frontline chemotherapy.

DETAILED DESCRIPTION:
Approximately two-thirds of patients with Hodgkin lymphoma (HL) can be cured with standard frontline chemotherapy with doxorubicin, bleomycin, vinblastine and dacarbazine (ABVD). The majority of new patients present in the second and third decade of life, but at least 25% of de novo cases are in patients older than 65. Elderly patients with HL display dismal outcomes for several reasons: the disease is implicitly more aggressive than in younger adults, with an advanced stage in at least two-thirds of cases and the presence of multiple risk factors for poor outcome (according to the International Prognostic Score). Moreover, patients may show impaired organ function that require chemotherapy dose reductions, treatment delays or drug withdrawal.

Given the difficulty of delivering of full treatment doses to elderly patients and to those with relevant medical comorbidities, there is a need for new and better tolerated agents in this context.

Given the difficulty of delivering of full treatment doses to elderly patients and to those with relevant medical comorbidities, there is a need for new and better tolerated agents in this context. Importantly, no single agent has received approval for this kind of patients, and drugs like gemcitabine and bendamustine - both active in relapsed patients with limited toxicity - have limitations in their prescription. The anti-CD30 immunoconjugate agent brentuximab vedotin (BV) applied in patients older than 60 years and considered unsuitable for frontline chemotherapy, yielded an overall response of 92%, with 73% of patients achieving a complete remission and a median duration of response of 9.1 months.

Immune checkpoint inhibitors, namely nivolumab and pembrolizumab, have been largely tested in patients with relapsed and refractory HL failing both autologous stem cell transplant and BV. Both agents display efficacy in this context, with significant rates of objective responses, which appear to be durable. Along with an acceptable safety profile, both agents have been approved in relapsed and refractory HL, providing a good treatment option for heavily pretreated patients. Tislelizumab (T, BGB-A317) is a humanized IgG4 mAb with high affinity and specificity for programmed cell death protein 1 (PD1), showing a superior antitumor activity compared to nivolumab in mice transplanted with human cancer cells and peripheral blood mononuclear cells. High response rates have been reported in Chinese HL patients who have failed or were ineligible to autologous transplantation, including a complete response rate of 61% and a partial response rate of 24%.

Investigators postulate that an induction based on single-agent tislelizumab can be a feasible chemo-free treatment strategy to be offered to patients with de novo HL who are unsuitable for a chemotherapy-based frontline approach.

The study also addresses biological evaluation of biomarkers in the tumor clone and in the microenvironment at baseline and their possible correlation with patients' outcome and responses.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of de novo classical Hodgkin Lymphoma (cHL). Note: Availability of either block or unstained slides plus stained slides used by the local pathologist to make diagnosis, and of all pathology reports is mandatory for the study to perform central pathology review for confirmation of cHL diagnosis and for biological biomarkers assessments. Central pathology confirmation is not required to start treatment;
* Patients >= 65 years ineligible for frontline standard chemotherapy (mainly due to medical comorbidities);
* Treatment naïve;
* Measurable disease defined as presence of both fluorodeoxyglucose-avid nodal involvement and at least one nodal target lesion measurable in two diameters (and at least 1.5 cm in its major diameter); • Indication for systemic treatment, i.e., all stages except IA without a large tumor burden, as radiotherapy is regarded curative in those patients;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) <= 2;
* Adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) > 109/L (without growth factor support within 7 days of ANC measurement), unless due to bone marrow involvement by lymphoma
  * Platelet > 50 x 109/L (without growth factor support or transfusion within 7 days of platelets measurement) , unless due to bone marrow involvement by lymphoma
  * Hemoglobin > 8 g/dL (prior transfusion is acceptable)
  * Creatinine clearance ≥ 30 ml/min (as estimated by the Cockcroft-Gault equation or as measured by nuclear medicine scan or 24-hour urine collection)
  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase, and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase ≤ 3.0 × upper limit of normal (ULN)
  * Serum total bilirubin < 1.5 × ULN (or < 3 x ULN in case of documented Gilbert's syndrome)
* Life expectancy ≥ 6 months;
* Men must agree to use effective contraception if sexually active. This applies for the time period between signing of the informed consent form and 4 months after last tislelizumab dose. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control method, e.g. vasectomy, use of condoms or complete sexual abstinence, when this is in line with the preferred and usual lifestyle of the subject.The use of condoms by male patients is required unless the female partner is permanently sterile. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods for the female partner) and withdrawal are not acceptable methods of contraception.
* Subject voluntarily signs and dates an informed consent form approved by an National Ethics Committee (NEC) prior to the initiation of any screening or study-specific procedures, indicating that they understand the purpose of and procedures required for the study and are willing to participate in it;
* Subject must be able to adhere to the study visit schedule and other protocol requirements, and to return to enrolling institution for follow-up (during the active monitoring phase of the study).

Exclusion Criteria:

* Nodular lymphocyte predominant HL;
* Any previous treatment (including radiation therapy) for HL;
* Any active autoimmune disease requiring systemic treatment (including disease-modifying agents, corticosteroids, immunosuppressants) in the past 2 years; Note: Patients with the following diseases are not excluded and may proceed to further screening: Type I diabetes under control; Hypothyroidism (provided it is managed with hormone replacement therapy only); Controlled celiac disease;
* Has known history of interstitial lung disease, non-infectious pneumonitis, pulmonary fibrosis, acute lung diseases or evidence of dyspnea at rest or pulse oximetry of < 92% while breathing room air;
* A history of previous exposure to anti-PD1, anti-PDL1 or anti-PDL2 or anti-CTLA-4 agents for any disease other than HL;
* Use of systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications ≤14 days from registration; Note: Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease;
* Known infection with HIV, human T-cell lymphotropic virus-1, -2; • Serologic status reflecting active hepatitis B defined as presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) (mandatory testing). Patients with occult or prior HBV infection (respectively defined as patient with HBsAg-/HBcAb+ and patients HBsAg+ with HBV DNA undetectable) are eligible, provided that they are willing to undergo prophylactic antiviral medication according to local standard of care. Patients who have protective titers of hepatitis B surface antibody (HBsAb) after vaccination are eligible;
* Presence of hepatitis C virus (HCV) antibody (mandatory HCV antibody serology testing). Patients with presence of HCV antibody are eligible only if PCR is negative for HCV RNA;
* Hypersensitivity to tislelizumab or any of its excipients;
* Active central nervous system (CNS) involvement or leptomeningeal metastases involvement;
* Evidence of other clinically significant uncontrolled and/or active systemic infection (viral, bacterial or fungal), including active ongoing infection from SARS-CoV-2;
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens;
* Major surgery within 4 weeks of the first dose of study drug;
* Vaccination with a live vaccine within 4 weeks prior to the first dose of study drug;
* Clinically significant cardiovascular disease including the following:

  * Myocardial infarction within 6 months before screening;
  * Unstable angina within 3 months before screening;
  * New York Heart Association Classification III or IV congestive heart failure;
  * History of clinically significant arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsade de pointes);
  * QTcF > 480 msecs based on Fridericia's formula;
  * History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place;
  * Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mm Hg and diastolic blood pressure > 105 mm Hg at screening;
* Significant history of neurologic, psychiatric, endocrinological, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent;
* Any history of other active malignancies within 3 years prior to study entry, with the exception of adequately treated in situ carcinoma of the cervix uterine, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, previous malignancy confined and surgically resected with curative intent;
* History of severe hypersensitivity reactions to other monoclonal antibodies;
* Concurrent participation in another therapeutic clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (CR + PR) | From treatment start up to about 24 months
  The primary endpoint of the study is the ORR (the sum of complete response (CR) and partial response (PR) rate).

SECONDARY OUTCOMES:
Duration of response (DoR) | Between +33 days after treatment start up to 66 months
  Time from first documented complete response according to Lugano and LYRIC criteria to disease relapse.
Progression-free survival (PFS) | From registration up to 66 months
  Time from registration to the earliest date of documentation of disease progression, relapse or death from any cause.
Overall survival (OS) | From registration up to 66 months
  Time from registration to death from any cause.
Disease free survival (DFS) | Between +33 days after treatment start up to 66 months
  Time from first documented complete response according to Lugano and LYRIC criteria to disease relapse or death as a result of lymphoma or acute toxicity of treatment.
Incidence and severity of adverse events occurred during therapy and up to 90 days after treatment and incidence and severity of serious adverse events occurred from the IC signed to the end of the study (LPLV) | From treatment start up to 66 months
  To evaluate the safety and tolerability of tislelizumab

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — Istituto di Ematologia "L. e A. Seràgnoli", AOU Policlinico S.Orsola-Malpighi, Bologna
Locations (10):
- Italy (10):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, S.C. Ematologia, Alessandria, IT
  - Divisione di Oncologia e dei Tumori immuto-correlati, Centro Di Riferimento Oncologico Di Aviano, Aviano
  - Istituto di Ematologia L. e A. Seràgnoli, AOU Policlinico S. Orsola-Malpighi, Bologna
  - SC Ematologia, Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Ematologia, Fondazione IRCCS Istituto Nazionale Dei Tumori, Milan
  - Unità di Ematologia e TMO - Unità Linfomi, Ospedale San Raffaele, Milan
  - Oncologia, IRCCS Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Oncoematologia, Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione, Azienda Ospealiero Universitaria Policlinico Umberto I, Roma
  - U.O di Oncologia Medica ed Ematologia, Humanitas Research Hospital, Rozzano